CLINICAL TRIAL: NCT02427958
Title: An Open Label, Multicenter Study to Assess the Safety and Efficacy of Leuprorelin in the Treatment of Central Precocious Puberty
Brief Title: A Study to Assess the Safety and Efficacy of Leuprorelin in Central Precocious Puberty in Chinese Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Leuprorelin-4001; U1111-1183-0353 (Registry Identifier: WHO); CTR20140148 (Registry Identifier: SFDA CTR)
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Central Precocious Puberty
Keywords: Drug Therapy
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Leuprorelin (Experimental): Participants with body weight greater than or equal to (>=) 20 kilogram (kg) will receive the recommended dose of leuprorelin 3.75 milligram (mg), injection, subcutaneously, once every 4 weeks for 96 weeks. Participants with body weight less than (<) 20 kg will receive leuprorelin 1.88 mg, injection, subcutaneously, once every 4 weeks for 96 weeks.
  Interventions: Drug: Leuprorelin

INTERVENTIONS:
Drug: Leuprorelin — Suspension for injection.
  Other Names: Enantone

SUMMARY:
The purpose of this study is to assess long-term safety and efficacy of leuprorelin in the treatment of Central Precocious Puberty (CPP).

DETAILED DESCRIPTION:
The drug in this study is called leuprorelin. It is administered as a 1 month subcutaneous depot injection. Leuprorelin is used to treat children who have CPP. This study will look at whether leuprorelin can stop early puberty in pre-pubertal children.

The study will enroll approximately 300 participants. Participants with body weight >=20 kg will receive the recommended dose of leuprorelin 3.75 mg subcutaneous injection every 4 weeks for 96 weeks. Participants with body weight <20 kg will receive recommended dose of 1.88 mg subcutaneous injection every 4 weeks for 96 weeks.

This trial will be conducted in China. The overall time to participate in this study is 104 weeks. Participants will make 11 visits to the clinic, and will be followed-up by the physician on a long-term basis until stable puberty is reached.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant and/or parent(s) or legal guardian are capable of understanding and complying with protocol requirements.
2. The participant or the participant's parent(s) or legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. Has onset of appearance of secondary sexual characteristic earlier than age 8.0 years in girls or earlier than 9.0 years in boys and the symptom is persistent, and has confirmed diagnosis of CPP.
4. Has basal luteinizing hormone (LH) level greater than (>) 5.0 international units per liter (IU/L) or peak LH >3.3 IU/L with LH/follicle-stimulating factor (FSH) >0.6 in stimulation test.
5. Has evidence of gonadal development evaluated by ultrasonography: ovarian volume >=1 milliliter (mL) with multiple follicles >=4 millimeter (mm) in any ovary or uterine enlargement in females or testicular volume >=4 mL in males.
6. Has advanced bone age (BA) >=1 year and BA is less than or equal to (<=) 11.5 years in females or <=12.5 years in males OR predicted adult height <150 centimeter (cm) in females or <160 cm in males OR standard deviation score (SDS) <-2 standard deviations (SD) OR rapid growth defined as growth of BA /growth of chronologic age >1. BA is determined by Greulich and Pyle standards or Tanner-Whitehouse 3 (TW3) standards at screening.
7. Has anticipated treatment duration of at least 2 year in investigator's judgment.
8. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 90 days after last dose.
9. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.
10. The female participant who, at the discretion of the investigator, is deemed to be of child bearing potential must provide negative urine pregnancy text at Day -1 or Day 1 prior to drug administration.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Has received gonadotropin-releasing hormone analog (GnRHa) treatment in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (example [eg], spouse, parent, child, sibling) or may consent under duress.
4. Has any findings in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of underlying disease that might interfere with the conduct of the trial.
5. Has any concomitant medical condition that, in the opinion of the investigator, may expose a participant to an unacceptable level of safety risk or that affects participant compliance.
6. Has any screening abnormal laboratory value that suggests a clinically significant underlying disease or condition that may prevent the participant from entering the study; or the participant has: creatinine >=1.5 milligram per deciliter (mg/dL), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) >2 times the upper limit of normal (ULN), or total bilirubin >2.0 mg/dL, with AST/ALT elevated above the limits of normal values.
7. Has a history or clinical manifestations of significant adrenal or thyroid diseases or intracranial tumor OR has a history of malignant disease.
8. Has a history of hypersensitivity or allergies to leuprorelin, or related compounds including any excipients of the compound.
9. Has a diagnosis of peripheral precocious puberty.
10. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the Screening Visit.
11. Participant or parent(s), at the discretion of the investigator, is unlikely to comply with the protocol or is unsuitable for any of other reason.
12. If female, the participant is of childbearing potential (eg, not sterilized).
13. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
14. If male, the participant intends to donate sperm during the course of this study or for 90 days thereafter.
15. Has participated in another clinical study and/or has received any investigational compound within 30 days prior to Screening.

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 307 (Actual)
Dates: Start 2015-08-07 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (9):
- China (9):
  - Beijing, Beijing Municipality
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nanjing, Jiangsu
  - Wuxi, Jiangsu
  - Nanchang, Jiangxi
  - Changchun, Jilin
  - Shanghai, Shanghai Municipality
  - Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Luo X, Hou L, Zhong Y, You C, Yang Y, Wu X, Li P, Zhou S, Qiu W, Zhang H, Liu Y, Qian Y, Luo F, Cheng R, Hu Y, Gong H, Wang Q, Xu Z, Du H, Lu F, Fu J, Chen X, Wang W, Guo Z. An open label, multicenter clinical trial that investigated the efficacy and safety of leuprorelin treatment of central precocious puberty in Chinese children. Medicine (Baltimore). 2021 Dec 23;100(51):e28158. doi: 10.1097/MD.0000000000028158. PMID 34941067

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 11 investigative sites in China from 07 August 2015 to 23 November 2018.
Pre-assignment Details: Chinese participants with central precocious puberty (CPP) were enrolled to receive leuprorelin as per body weight.
Groups:
- Leuprorelin: Participants with body weight greater than or equal to (>=) 20 kilogram (kg) received the recommended initial dose of leuprorelin 3.75 milligram (mg), injection, subcutaneously, once every 4 weeks for 96 weeks. Participants with body weight less than (<) 20 kg received leuprorelin 1.88 mg, injection, subcutaneously, once every 4 weeks for 96 weeks. The dose was adjusted based on participant's condition and investigator's judgment in alignment with the product label in China.
Period: Overall Study
Arm/Group | Leuprorelin
Started | 307
Completed | 283
Not Completed | 24
Not completed — Pretreatment Event (PTE) or AE | 3
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 14
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Leuprorelin
Number analyzed (Participants) | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.03 (0.935)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 305
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 307
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 307
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 133.68 (7.108)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 30.44 (5.346)
Weight Categories [Count of Participants; unit: Participants]
  <20 kg | 5
  >=20 kg | 302
Age at date of diagnosis of CPP [Mean (Standard Deviation); unit: years] — Population: Number of participants for whom Age at date of diagnosis of CPP data was available in baseline characteristics was 296.
  years
    number analyzed (Participants) | 296
    (all) | 7.95 (0.982)
Tanner Staging Evaluation: Breast (Female) and Genitals (Male) [Count of Participants; unit: Participants] — Tanner assessment score was used to document the stage of development of puberty by assessing the secondary sexual characteristics. Female pubertal development staged by breast size; male pubertal development staged by size of the genitalia. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
  Participants
    Stage 1 | 3
    Stage 2 | 172
    Stage 3 | 120
    Stage 4 | 11
    Stage 5 | 1
Tanner Staging Evaluation: Pubic Hair [Count of Participants; unit: Participants] — Tanner assessment score was used to document the stage of development of puberty by assessing the secondary sexual characteristics (pubic hair) in male and females. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size).
  Participants
    Stage 1 | 266
    Stage 2 | 31
    Stage 3 | 9
    Stage 4 | 0
    Stage 5 | 1
Peak Stimulated Luteinizing Hormone (LH) [Mean (Standard Deviation); unit: unit per liter (U/L)] | 20.664 (18.1982)
Peak Stimulated Follicle-stimulating Hormone (FSH) [Mean (Standard Deviation); unit: U/L] | 14.992 (6.7343)
Bone Age/Chronological Age [Mean (Standard Deviation); unit: ratio] — Population: Number of participants for whom bone age/chronological age data was available in baseline characteristics was 304.
  ratio
    number analyzed (Participants) | 304
    (all) | 1.26 (0.139)
Bone Mineral Density [Mean (Standard Deviation); unit: gram per square centimeter (g/cm^2)] — Population: Number of participants for whom bone mineral density data was available in baseline characteristics was 182.
  gram per square centimeter (g/cm^2)
    number analyzed (Participants) | 182
    (all) | 0.4791 (0.2142)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Time Frame: Day 1 up to Week 100
Population: The safety analysis set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Leuprorelin
Number analyzed (Participants) | 307
participants | 252

2. Secondary Outcome: Percentage of Participants With Regression or no Progression in Tanner Staging at Week 96
Description: Tanner assessment score was used to document the stage of development of puberty through the assessment of secondary sexual characteristics. Female pubertal development staged by pubic hair development and breast size; male pubertal development staged by size of the genitalia and development of pubic hair. Rated in 5 stages: stage 1 (no development) to 5 (adult-like development in quantity and size). Regression or no progression was defined as negative change (improvement) or no change in Tanner score at Week 96 compared to baseline.
Time Frame: Week 96
Population: The full analysis set included all enrolled participants who received at least 1 dose of study drug. The full analysis set where data at specified time points was available.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprorelin
Number analyzed (Participants) | 307
percentage of participants
  Female: number analyzed (Participants) | 238
  Female | 83.5 [78.68 to 87.62]
  Male: number analyzed (Participants) | 2
  Male | 0 [0 to 84.19]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and no more than 30 days (Week 100) after the last dose of study drug
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Leuprorelin
All-Cause Mortality (participants affected / at risk) | 0/307
Serious Adverse Events (participants affected / at risk) | 12/307
Other Adverse Events (participants affected / at risk) | 189/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin (N=307)
Pneumonia (Infections and infestations) | 4
Pneumonia mycoplasmal (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Chronic tonsillitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 1
Epiphyseal injury (Injury, poisoning and procedural complications) | 1
Peripheral nerve injury (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin (N=307)
Upper respiratory tract infection (Infections and infestations) | 118
Cough (Respiratory, thoracic and mediastinal disorders) | 51
Pyrexia (General disorders) | 45
Nasopharyngitis (Infections and infestations) | 35
Bronchitis (Infections and infestations) | 34
Tonsillitis (Infections and infestations) | 19
Pharyngitis (Infections and infestations) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2015-12-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT02427958/Prot_001.pdf
  • Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT02427958/SAP_000.pdf